CLINICAL TRIAL: NCT05394272
Title: Efficacy of Energy Therapy in the Management of Chronic Pain and Associated Medical Condition in Children and Adolescents.
Brief Title: Efficacy of Energy Therapy in the Management of Chronic Pain Medical Condition in Children and Adolescents.
Acronym: ET&CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KCH22-058
Record Dates: First submitted 2022-05-04; First posted 2022-05-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn Disease; Chronic Pancreatitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: Longitudinal, experimental qualitative and quantitative research project. Non-pharmacological, non- invasive, natural complementary therapy.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of Energy Therapy - Pranic Healing with chronic pain (Experimental): Energy therapy - Pranic Healing to be applied for 8 weeks weekly and 3 times 4 weeks apart for relief of chronic pain
  Interventions: Other: Energy Therapy - Pranic Healing
- Efficacy of Energy Therapy - Pranic Healing - with linked medical condition (Experimental): Energy Therapy - Pranic Healing protocol for linked medical condition applied for 8 weeks weekly and 3 times 4 weeks apart , relevant BT/Urine sample /stool sample 4 weeks apart to evaluate changes.
  Interventions: Other: Energy Therapy - Pranic Healing

INTERVENTIONS:
Other: Energy Therapy - Pranic Healing — Energy therapy - Non invasive non touch and non pharmacological - 100% natural complementary therapy

SUMMARY:
Paediatric and adolescent patients with chronic pain associated with their medical condition will be invited to participate in this study. Most patients for this study will be recruited from gastroenterology and hepatology clinics at KCH. Therefore the rationale for the study is primarily with consideration of each of these medical conditions all with the common symptom of chronic pain. Inflammatory bowel disease disorders(IBD), such as Crohn's Disease and Ulcerative Colitis, disorders of gut-brain interaction (DGBI) all experience chronic pain. however children with DGBI do not have an underlying specific lesion causing the pain. The chronic pain is the disease. In addition to this Chronic pancreatitis in children and adolescents can cause severe pain.

All of these groups of patients suffer with chronic pain and this can result in failure to thrive and have a negative impact on quality of life.

There is a need for further development of a non - pharmacological approach to support these patients with their symptoms of pain and in turn improve quality of life.

This study is designed to evaluate the benefits of a complementary natural therapy for paediatric and adolescent patients registered at King's College Hospital, with a diagnosis of a disease or disorder with associated symptoms of chronic pain. The age group is 5-18 years old.

The therapy to be evaluated is an energy therapy (Pranic Healing). This therapy is non -invasive, non- touch, non- pharmacological and natural. The study will assess the benefits these patients experience with their symptoms of pain after 8 weeks of weekly energy therapy sessions each session is 30 minutes and 3 visits each 4 weeks apart.

Qualitative and Quantitative data will be collected and evaluated.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study is to evaluate how effective a complementary therapy, Energy Therapy (Pranic Healing) is for children and adolescents that experience chronic pain.

Secondary Objective:

To evaluate efficacy of this energy therapy in reduction in clinical symptoms/pathology associated with the child's / adolescent's medical condition causing the chronic pain.

Longitudinal, experimental qualitative and quantitative research project. Non-pharmacological, non- invasive, natural complementary therapy.

The study is a controlled trial without randomisation experimental, longitudinal study designed to evaluate the efficacy of a non - pharmacological complementary therapies for children and adolescents with chronic.All participants are patients at King' College Hospital.

Recruitment

The initial recruitment for the study will be for patients from Gastroenterology and hepatology clinics at King's College Hospital. Patients with chronic pain with other medical conditions will be recruited as study progresses.

All families will be contacted by the medical care team or via the patient database by post/email with the PIL/PIS and ET information booklet (age appropriate).

Families will be contacted via email/ telephone, those interested in participation will be invited to an informal information session virtually or face to face.

The PIS will be discussed, any concerns regarding the study will be clarified. Parents will be asked to give informed consent if they would like their child to participate.

All participants will continue with their routine medical care and treatment at King's College Hospital.

Baseline Characteristics

To be collected prior to the intervention.

Pain -Visual Analogue Scale P-VAS - to be completed for 10 days prior to first session and daily for the duration of the study

Paediatric Ulcerative Colitis Activity Index (PUCAI) questionnaire- to be completed prior to the first session, subsequently every 4 weeks for the duration of the study for those patients with Ulcerative Colitis.

Paediatric Crohn's Disease Activity Index (PCDAI) questionnaire -to be completed prior to the first session subsequently every 4 weeks for the duration of the study for those patients with Crohn's Disease.

Faecal Calprotectin (FCP) - IBD PATIENTS will give a stool sample for a FCP test prior to their first session. Parents may bring the sample with them on the first appointment.

FCP samples will then be collected every 4 weeks for the duration of the study for patients with IBD.

Amylase (Blood test /Urine sample) BT/US Baseline level from last sample - patient records, collect sample at 4 weeks 8 weeks and 20 weeks (CP patients and pts where blood test routinely collected to evaluate clinical /physical symptoms).

Height and Weight (H&W) will be recorded at the first visit and every 4 weeks for the duration of the study for all patients.

Medication - a table recording medication dosage and frequency for abdominal pain will be requested to be completed for 10 days prior to the first session and every day throughout the study.

Journal - A diary will be given to patients /parents for young children,10 days prior to the study and for completion logging any changes through the study with pain associated with

Inflammatory Bowel Disease ( Ulcerative Colitis and Crohn's Disease) and Disorders of Gut- Brain Interaction and Chronic Pancreatitis and other medical conditions with manifestations of chronic pain 100

1. Recruitment process via referral from medical care team and patient database (registered paediatric and adolescent patients with chronic pain linked with medical condition at KCH)
2. Post/email PIS/PIL age appropriate information booklet
3. Informal information session / patient screening
4. Parent /adolescent giving consent if wishing to participate
5. Letter to GP informing of participation in study.
6. Letter to school /employer with dates and times of appointments where appropriate and requested.
7. 10 days prior to first session P-VAS completed daily Medication table for pain daily Journal
8. First appointment for Energy Therapy- prior to session PUCAI or PCDAI for IBD participants. Collection of FCP/BT/ US sample, if baseline not available in patient records. H&W.
9. Daily completion of P-VAS/medication for pain and journal
10. Weekly visits for 8 weeks - 30 minutes each visit
11. 4 weeks stage PUCAI/PCDAI/FCP/BT/US/H&W to be collected.
12. 8 week stage PUCAI/PCDAI/ H&W /FCP/BT/US to be collected.
13. Energy Therapy sessions to be every 4 weeks for 3 months. For the 3 visits PUCAI/PCDAI/H&W/FCP/BT/US For the final visit BT/US collection in addition.

22 weeks

Inclusion Criteria:

Registered Paediatric patient at King's College Hospital 5-18years of age Male and Female Diagnosis of medical condition with associated chronic pain Symptoms of Pain

Exclusion Criteria

Under 5 years old and older than 18 years old

No symptoms of pain

ELIGIBILITY:
Inclusion Criteria:

* Registered patients at King's College Hospital Male and Female 5-18 years old Symptoms of chronic pain associated with medical condition

Exclusion Criteria:

* Under 5 years of age and older than 18 years No symptoms of pain

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
P-VAS validated questionnaire | 20 weeks
  reduction in symptoms of chronic pain with Energy therapy

SECONDARY OUTCOMES:
stool samples/urine samples and blood tests | Patient will have 8 weeks of treatment - 1 x week and 3 reviews 4 weeks apart
  stool samples - faecal calprotectin
  Faecal calprotectin

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No